CLINICAL TRIAL: NCT05524766
Title: Evaluation of Safety and Efficacy of the BTL-785F Device for Non-invasive Facial Rejuvenation in Patients Injected With Botulinum Toxin
Brief Title: BTL-785F Device for Non-invasive Facial Rejuvenation in Patients Injected With Botulinum Toxin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS1100
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BTL-785-7 Treatment (Experimental): Subjects will be enrolled for an active treatment with BTL-785F device (BTL-785-7 applicator) for improvement of overall facial appearance and muscle tone in patients injected with botulinum toxin.
  Interventions: Device: BTL-785-7 Treatment
- Control (No Intervention): Two (2) patients will be enrolled in the control group study and will not receive any treatment. Following the completion of the investigation, the control group patients will be offered the same treatment course as the active group.

INTERVENTIONS:
Device: BTL-785-7 Treatment — Treatment with BTL-785F device (BTL-785-7 applicator) for improvement of overall facial appearance and muscle tone in patients injected with botulinum toxin.
  Arms: BTL-785-7 Treatment

SUMMARY:
This study will evaluate the clinical safety and the efficacy of the BTL-785F system equipped with the BTL-785-7 applicator for non-invasive facial treatment in patients injected with botulinum toxin. The aim is to investigate the improvement of overall facial appearance and muscle tone.

DETAILED DESCRIPTION:
This study is a single-site, open-label, interventional study. The subjects will be enrolled and assigned into two experimental study arms (active and control group).

At the baseline visit health status will be assessed and, if needed, additional tests will be performed. Inclusion and exclusion criteria will be verified and informed consent will be signed.

The treatment administration phase (only for the active group) consists of four (4) treatment visits, delivered 5-10 days apart.

Safety measures will include documentation of adverse events (AE) including the subject's experience of pain or discomfort after the procedure. Occurrence of AE's will be checked immediately after the first treatment visit, prior/post to the every other procedure and at the follow-ups.

Subjects will undergo two follow-up visits scheduled at 1 month and 3 months after the final treatment (the control group will not receive any treatment).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for reduction of wrinkles and overall aesthetic improvement of the face
* Subjects injected with type A botulinum toxin for facial wrinkles improvement in the past month, but no sooner than 1 week
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Electroanalgesia without exact diagnosis of pain etiology
* Serious psychopathological disorders (such as schizophrenia)
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Facial Appearance Change | 5 months
  Three evaluators will evaluate facial appearance according to the Global Aesthetic Improvement Scale (GAIS) using the photographs taken at the baseline, last therapy visit and both follow-up visits. Each evaluator will be asked to assign a score to a set of photographs. The GAIS is a clinically validated assessment tool used to assess overall aesthetic improvement such as facelift on a scale from -1 through 3, where the higher score is considered better.
  The baseline and post-treatment scores will be compared. If applicable, the statistical significance of obtained results will be analyzed in Microsoft Excel spreadsheet software. The level of significance (α) will be set as 5%.

SECONDARY OUTCOMES:
Facial expression assessment | 5 months
  Short facial expression records will be taken for evaluating the level of change in the facial expression. The patients will be required to perform happy, angry, and surprised expressions. The video of patients facial expressions will be taken at baseline, after the treatment, and at all follow-up visits. These records will be also evaluated with GAIS scoring. The GAIS is a clinically validated assessment tool used to assess overall aesthetic improvement such as facelift on a scale from -1 through 3, where the higher score is considered better.
Therapy Comfort | 5 months
  The 7-point Likert scale Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. Pain sensation will be rated by the subjects from 0 (no pain) to 10 (worst possible pain).
Subject Satisfaction | 5 months
  The 7-point Likert scale Subject Satisfaction Questionnaire will be used for evaluating the satisfaction. The Subject Satisfaction Questionnaire will be given to subjects after the last therapy, at 1-month and 3-month follow-up. The answers to the questions related to the subjects' overall skin and face appearance will vary from "strongly agree" to "strongly disagree".

CONTACTS AND LOCATIONS:
Locations (1):
- Refresh Dermatology, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No